CLINICAL TRIAL: NCT01461733
Title: Atrial Fibrillation WITHOUT Hemodynamic Stability
Brief Title: Atrial Fibrillation Without Hemodynamic Instability in the Intensive Care Unit
Acronym: AFIB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, S. Kanji, MD, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA5936 Heart and Stroke; OHREB Protocol # 2006430-01 (Other Grant/Funding Number: heart and stroke foundation of ON)
Record Dates: First submitted 2010-08-19; First posted 2011-10-28 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; amiodarone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- amiodarone (Experimental): standard dose amiodarone
  Interventions: Drug: amiodarone
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: amiodarone — standard dose amiodarone
  Other Names: non applicable
  Arms: amiodarone
Drug: Placebo — placebo delivered blinded
  Arms: placebo

SUMMARY:
Atrial fibrillation (AF) is an abnormal heart rhythm that is common among patients who are admitted to an intensive care unit (ICU) of a hospital. It is usually a transient occurrence that resolves as the patient recovers from their underlying condition. However, patients who develop AF can present with a very rapid heart rate that in some cases can put stress on the heart which can lead to life threatening heart attacks, low blood pressure or breathing problems. Not all patients with AF will have unstable heart function but those who have rapid heart rates can worsen quickly. The goals of treatment for AF with a rapid heart rate but no unstable heart function are two fold. Patients can be treated by controlling the heart rate and/or by attempting to convert the AF to a normal heart rhythm. The heart rate can be controlled by medication and the AF can be converted by either electrical cardioversion (an electric shock that jump-starts the heart) or medication. Currently it is unknown if the goal of treatment should be to simply control the heart rate and wait for the patient to spontaneously convert to a normal heart rhythm or convert the AF with medication for patients who only have the rapid heart rate.

The objective of this project is to conduct a pilot study to determine if it would be feasible to conduct a larger definitive trial that would answer the following question: Should the goal of treatment be to control the rapid heart rate or resolve the abnormal heart rhythm in patients with AF who have a rapid heart rate without unstable heart function.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* new onset afib

Exclusion Criteria:

* hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salmaan Kanji, MD, Principal Investigator — Ottawa Hospital Research Institute

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amiodarone | Placebo
Started | 12 | 12
Completed | 8 | 8
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amiodarone | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (17) | 61 (17) | 65 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Conversion From Atrial Fibrillation to Sinus Rhythm
Description: Conversion rates measured during ICU stay only. Average duration of ICU stay is 7 days.
Time Frame: From randomization to conversion or ICU discharge up to 100 months.
Measure: Number; unit: participants
Arm/Group | Amiodarone | Placebo
Number analyzed (Participants) | 8 | 8
participants | 8 | 5

ADVERSE EVENTS:
Arm/Group | Amiodarone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes